CLINICAL TRIAL: NCT05138627
Title: The Effect of Oral Cryotherapy on Anticipatory, Acute and Late Nausea and Vomiting in Breast Cancer Patients Receiving Adjuvant Chemotherapy Treatment
Brief Title: The Effect of Oral Cryotherapy on Anticipatory, Acute and Late Nausea and Vomiting in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berna KURT (Other)
Responsible Party: Sponsor-Investigator, Berna KURT, Principal Investigator, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA-20007
Record Dates: First submitted 2021-10-19; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: nursing; nausea vomiting; randomized controlled trial; oral cryotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): 1. Teaching of oral cryotherapy by the investigator in the hospital,
  2. Implementation of oral cryotherapy accompanied by the investigator in the hospital
  3. Individual application of oral cryotherapy at home by patients
  Interventions: Other: oral cryotherapy
- control (No Intervention): Routine procedures in the clinic were performed on the first course (day 0) when the patients came to receive adjuvant chemotherapy and every 21 days thereafter, and oral cryotherapy was not applied to the patients. Before applying the first adjuvant chemotherapy, Nausea Vomiting Training and Guide was given to have equal conditions with the patients in the intervention groups.

INTERVENTIONS:
Other: oral cryotherapy — Ice application protocol developed by the researcher by scanning the literature was prepared by taking the opinions of 5 faculty members who are experts in their fields. Also, the chamber of physics engineers and the chamber of chemical engineers' opinion was taken for the necessary corrections or improvements regarding the chemical/physical structure of the ice and the method applied. In the content of the protocol, materials, preparation before intraoral ice application (written and visual), steps of intraoral ice application (written and visual), termination of intraoral ice application, recording of intraoral ice application, and situations to be considered are explained in detail respectively.
  Arms: intervention

SUMMARY:
The purpose of this randomized controlled, statistical blind study that has an intervention control group was to determine the effect of oral cryotherapy on anticipatory, acute, and late nausea and vomiting of breast cancer patients receiving adjuvant chemotherapy. The study was carried out between July 2020-May 2021 in the Unit of the Medical Oncology Department of University of Health Sciences Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital. The study sample consisted of 54 breast cancer patients. 26 patients belonged to the intervention group and 28 to the control group. They were stratified based on their ages and body surface areas and were planned to receive chemotherapy for four cycles. The Oral Cryotherapy Protocol; developed by the researcher was made by obtaining opinions of five academic members and physics engineers and chemical engineers. Nausea and vomiting training guide and education was given to all patients in the study to avoid discrimination. The intervention group of the study applied oral cryotherapy with the researcher when they came to the hospital for the treatment and at home. No procedure outside of the routine treatment was performed on patients in the control group. Data in the study were collected through the Patient Information Form, the Rhodes Index of Nausea Vomiting and Retching (RINVR), and the EORTC QLQ-C30 Life Quality Index. The effect of oral cryotherapy was measured by the RINVR by contacting the patients every day for the first week during four cycles. EORTC QLQ-C30 and RINVR were conducted on patients when they came to the hospital throughout their cycles.

DETAILED DESCRIPTION:
Nausea-vomiting (80%) is the leading symptom associated with chemotherapy. The chemotherapeutic regimen's emetogenicity is effective in the emergence of chemotherapy-induced nausea-vomiting (CINV). In CINV, centers such as the cerebral cortex and the gastrointestinal tract stimulated the Chemoreceptor Trigger Zone (CTZ). Cytotoxic drugs can easily reach the CTZ. Various emetogenic cause serotonin release from enterochromaffin cells in the gastrointestinal tract. Serotonin stimulates CTZ in the central nervous system, and emesis develops. Despite the antiemetic drugs given to prevent the side effects of chemotherapy drugs, 60% of patients experience nausea and vomiting. Adriamycin Cyclophosphamide (AC) chemotherapy agents often cause nausea and vomiting between 1-7th days after the treatment. When CINV cannot be controlled effectively and adequately, anticipatory nausea and vomiting develop, especially within 24 hours before chemotherapy treatment, and a learned reflex mechanism occurs. It is stated that uncontrolled anticipatory nausea and vomiting in adult patients triggers acute and late nausea and vomiting. It is indicated that approximately 70% of the patients who received chemotherapy treatment between the first and fifth days experienced vomiting at least once, and 80% of the patients experienced nausea at least once.

The guideline for the prevention and management of nausea-vomiting published by the Oncology Nursing Society (ONS) states that the use of non-pharmacological approaches together with pharmacological methods may be appropriate. One of the nonpharmacological applications recommended in the management of chemotherapy-related symptoms is oral cryotherapy. Cryotherapy is the process of cooling the tissues by utilizing the effect of pieces of ice. Cryotherapy causes local vasoconstriction when used in treatment with intravenously administered chemotherapy agents. The local effect of ice application in preventing muscle damage is that it causes vasoconstriction in blood and lymph vessels, reducing the inflammatory response and activation of some proteins. The most important neuroreceptors in the formation of the emetic response are serotonin, substance-P, dopamine, acetylcholine, corticosteroid, and histamine. The most important neurotransmitters are dopamine, serotonin, and substance-P. Substance-P stimulates cholinergic neurons, causing vasodilation, increased secretion, and smooth muscle contraction. This way, it triggers vomiting by stimulating the CTZ.

ELIGIBILITY:
The inclusion criteria were as follows;

* Between the ages of 18- 65
* Open to communication and cooperation, literate
* Knowing about their diagnosis
* Diagnosed with breast cancer for the first time
* Adjuvant chemotherapy protocol planned for the first time
* Receiving AC Protocol as chemotherapy protocol
* Who did not receive radiotherapy treatment before adjuvant chemotherapy
* Who does not have COPD, AMI, CHF, CRF, Gastrointestinal, Neurological, Metabolic, pregnancy and non-DM
* Who did not use a non-pharmacological method for nausea-vomiting
* Who received standard antiemetic therapy in accordance with the AC protocol
* Who does not have metastasis
* Who does not have thrombocytopenia
* Who has Stage I and Stage II breast cancer
* Who is not treated for psychiatric and/or depression
* Consisted of female patients who were willing and voluntarily to participate in the study.

The exclusion criteria were as follows;

* Treatment delayed at least two times in a row
* Unreachable through phone calls
* Changed treatment regimen/drugs
* Patients who stopped participating in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 54 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Rhodes Index of Nausea Vomiting and Retching (RINVR) | during four cycles of chemotherapy (each cycle is 21 days)
  The scale has three sub-dimensions as symptom experience, symptom occurrence, and symptom distress.

SECONDARY OUTCOMES:
EORTC QLQ-C30 Life Quality Index (EORTC QLQ-C30) | during four cycles of chemotherapy (each cycle is 21 days)
  The scale consists of three sub-dimensions as general well-being, functional difficulties, and symptom control.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Çakmak Öksüzoğlu, Professor, Study Director — bernacolakoglu85@gmail.com
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)